CLINICAL TRIAL: NCT04554589
Title: The Off Label Use of Glycopyrrolate in the Adults Intensive Care Unit.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, ICU consultant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000-0002-141
Record Dates: First submitted 2020-05-10; First posted 2020-09-18 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Effect of Drugs
MeSH Terms: interventions — Glycopyrrolate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- intervention group (Active Comparator): receive Glycopyrrolate at dose of 0.2 mg IV every 8 hours daily .
  Interventions: Drug: Glycopyrrolate 0.2 MG
- placebo group (Placebo Comparator): receive normal saline 2 ml IV every 8 hours daily .
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Glycopyrrolate 0.2 MG — injections
  Other Names: Glycopyrronium Injection
  Arms: intervention group
Drug: normal saline — normal saline
  Arms: placebo group

SUMMARY:
Tracheostomized patients in the ICU can have excessive tracheal secretions due to various causes as hyperactive airway, irritation of the mucus producing cells and inhibition of the ciliary functions. Excessive secretions will necessitate frequent suctions which carries the risk of tracheostomy tube obstruction if not managed properly. Excessive tracheal secretions may prolong the ICU stay, increase the nurses workload and increase patients morbidity and mortality.

This clinical trial hypothesizes that the use of glycopyrrolate may decrease the tracheal secretions and hence avoid such complications.

DETAILED DESCRIPTION:
Patients fulfilling the inclusion criteria will be randomly assigned into one of 2 groups:

Group G (Intervention group): Patients will receive Glycopyrrolate 0.2 mg IV every 8 hours.

Group C (Control group): Patients will receive 2 mL Normal saline every 8 hours.

Both injections will be labelled as drug A and drug B in the satellite pharmacy .

Both the attending physician, nurse and data collector will be blinded to the injection given.

Measurements data will be collected and recorded daily in the pre-prepared CRF during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years old.
2. Patients who are admitted to ICU for more than 72 hours.
3. Patients who have tracheostomy tubes with reported frequent need for suction of the tracheostomy tube secretions more than once every 4 hours.

Exclusion Criteria:

1. Patients who have evidence of lower respiratory tract infections and have positive cultures from the tracheal aspirate.
2. Patients who have known sensitivity to Glycopyrrolate.
3. Patients who have tachycardia (heart rate above 120 Beats/minute) or known to have tachyarrhythmiase.g atrial fibrillation.
4. Patients with mitral stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
Number of suctions per day | 6 days
  Number of suctions per day

SECONDARY OUTCOMES:
The duration of ICU days | 90 days
  the total days the patient will spend in ICU
Fio2 | 6 days
  Fio2 on mechanical ventilation every 4 hours daily
Mean airway pressure | 6 days
  Mean airway pressure will be recorded every 4 hours on the mechanical ventilator
Positive end expiatory pressure PEEP | 6 days
  PEEP will be recorded every 4 hours on the mechanical ventilator
The duration of mechanical ventilation days | 90 days
  Total days spent on mechanical ventilation
Side effects of Glycopyrrolate | 6 days
  Episodes of tachycardia if heart rate reach 120 beats / minute
Fluid intake | 6 days
  Fluid balance calculated daily
Total leukocyte count | 6 days
  Total leukocyte count daily

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abosamak, MD, Principal Investigator — health care provider
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data sharing will be participated after clinical trial registration complete.